CLINICAL TRIAL: NCT03901118
Title: A Multi-center, Phase Ⅱ Clinical Trial of Chiauranib Plus Chemotherapy in Relapsed/Refractory Ovarian Cancer
Brief Title: Chiauranib in Combination With Chemotherapy in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR201
Record Dates: First submitted 2019-03-29; First posted 2019-04-03 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer, relapsed or refractory; chiauranib, chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — chiauranib; Etoposide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chiauranib plus etoposide (Experimental): Patients receive the combined treatment of chiauranib plus etoposide, 28 days for a cycle, 6 cycles at most. In the pilot trial, Chiauranib is given orally, 25mg once daily. After patients finish the blood collection for pharmacokinetics(PK), and if the efficacy and safety are acceptable, Chiauranib is given orally, 50mg once daily. Etoposide is given orally, 50mg once daily for 21 days, 7 days off, in the pilot and formal study. After 6 cycles combined treatment, patients enter the single agent therapy of chiauranib.
  Interventions: Drug: chiauranib; Drug: etoposide
- chiauranib plus paclitaxel (Experimental): Patients receive the combined treatment of chiauranib plus paclitaxel, 21 days for a cycle, 6 cycles at most. In the pilot trial, Chiauranib is given orally, 25mg once daily. After patients finish the blood collection for pharmacokinetics(PK), and if the efficacy and safety are acceptable, Chiauranib is given orally, 50mg once daily. Paclitaxel is given in intravenous infusion on Day 1, 8 and 15, in the pilot and formal study. After 6 cycles combined treatment, patients enter the single agent therapy of chiauranib.
  Interventions: Drug: chiauranib; Drug: paclitaxel

INTERVENTIONS:
Drug: chiauranib — in the phase of pilot trial, 25mg orally once daily; in the formal phase, 50mg orally once daily
  Other Names: CS2164
Drug: etoposide — 50mg orally once daily for 21 days, 7 days off, every 28 days for a cycle, 6 cycles at most
  Other Names: Lastet
  Arms: chiauranib plus etoposide
Drug: paclitaxel — 60mg/m2, i.v infusion on day 1, 8 and 15, every 21 days for a cycle, 6 cycles at most
  Other Names: Anzatax
  Arms: chiauranib plus paclitaxel

SUMMARY:
This clinical trial will evaluate the efficacy and safety of chiauranib added to chemotherapy in patients with relapsed or refractory ovarian cancer, in the meantime, explore the pharmacokinetics characteristic after the combined treatment.

DETAILED DESCRIPTION:
This clinical trial will evaluate the efficacy and safety include adverse events, vital signs, laboratory tests, etc., of chiauranib added to chemotherapy (Paclitaxel/Etoposide) in patients with relapsed or refractory epithelial ovarian, fallopian tube or primary peritoneal cancer, in the meantime, explore the pharmacokinetics characteristic after the combined treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged ≥ 18 yrs and ≤70 yrs;
2. Histological or cytological confirmation of epithelial ovarian cancer, carcinoma tube, or primary peritoneal carcinoma.
3. Patients with platinum-resistant or platinum-refractory ovarian cancer,

   1. platinum-resistant disease (disease progression within 6 months of the last receipt of platinum-based chemotherapy);
   2. platinum-refractory disease (disease progression during the period of platinum-based chemotherapy);
   3. patients are platinum-sensitive for the first time, then disease progression within 6 months of the last receipt of platinum-based chemotherapy.
4. Patients have received at least 1 platinum containing chemotherapy (at least 4 cycles), the disease has progressed or relapsed no more than 2 different chemotherapy regimens.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. At least 1 lesion can be accurately measured, as defined by RECIST1.1.
7. The time for participants received anti-cancer therapy (including chemotherapy, radiotherapy, immunotherapy and surgical therapy, et al) should be more than 4 weeks before enrollment; The time for participants received mitomycin chemotherapy should be more than 6 weeks before enrollment.
8. Laboratory criteria are as follows:

   1. Complete blood count: hemoglobin (Hb) ≥90g/L ; absolute neutrophil count (ANC) ≥1.5×109/L ; platelets ≥90×109/L;
   2. Biochemistry test: serum creatinine(cr) <1.5×ULN; total bilirubin<1.5×ULN; alanine aminotransferase(ALT) ,aspartate aminotransferase(AST)≤2.5×ULN; (ALT,AST≦5×ULN if liver involved) ;
   3. Coagulation test: International Normalized Ratio (INR) < 1.5.
9. Life expectancy of at least 3 months.
10. Willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with prior invasive malignancies in the past five years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ;
2. Patients with allergic to Chiauranib, Etoposide and Paclitaxel;
3. Patients received vascular endothelial growth factor(VEGF)/vascular endothelial growth factor receptor(VEGFR) inhibitor, like Apatinib, Anlotinib, Fruquintinib, Bevacizumab, etc., or Aurora kinase inhibitors;
4. Patients received Etoposide therapy;
5. Patients received weekly Paclitaxel therapy ;
6. Clinical evidence of central nervous system involvement;
7. Have uncontrolled or significant cardiovascular disease, including:

   1. Congestive heart failure, unstable angina pectoris, myocardial infarction within 6 months prior to study entry; arrhythmia, or Left Ventricular Ejection Fraction (LVEF) < 50% requiring treatment with agents during screening stage.
   2. primary cardiomyopathy(dilated cardiomyopathy, hypertrophic cardiomyocyte, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, et,al)
   3. History of significant QT interval prolongation, or Corrected QT Interval (QTc) > 470 ms prior to study entry
   4. Symptomatic coronary heart disease requiring treatment with agents
   5. Uncontrolled hypertension (≥ 140/90 mmHg) by single agent.
8. Have active bleeding current thrombotic disease, patients with bleeding potential ,or receiving anticoagulation therapy; within 2 months prior to screening;
9. Proteinuria positive (≥1g/24h).
10. History of deep vein thrombosis or pulmonary embolism;
11. Have unsolved toxicities (> grade 1) from prior anti-cancer therapy;
12. Have clinical significant gastrointestinal abnormality, e.g., unable to swallow, chronic diarrhea, ileus, that would impair the ingestion, transportation or absorption of oral agents, or patients undergone gastrectomy;
13. History of organ transplantation;
14. Major surgery within 6 weeks and minor surgery within 2 weeks prior to screening;
15. Serologically positive for HIV, hepatitis B or C, or other serious infectious diseases (positive infectious diseases refer to that needed systemic therapy; HIV, hepatitis B or C: qualitative detection priority, quantitative detection if needed).
16. History of interstitial lung disease (ILD).
17. Any mental or cognitive disorder, that would impair the ability to understand the informed consent document or the operation and compliance of study;
18. Candidate with drug and alcohol abuse (alcohol abuse: alcohol consumption is no more than 5040ml beer or 2100ml wine or 630ml strong wine with alcohol content tops out at 40 percent each week).
19. Patients participated in other clinical trials in 4 weeks before enrollment, or washout period less than 5 half-life after received other clinical trial drugs (whichever is the longest);
20. Participants of reproductive potential not willing to use adequate contraceptive measures for the duration of the study (both male and female participants).Pregnant or breastfeeding women. Female participants must have a negative urinary or serum pregnancy test when done or have evidence of post-menopausal status (Defined as absence of menstruation for greater than 12 months, bilateral oophorectomy or hysterectomy).
21. Any other condition which is inappropriate for the study in the opinion of the investigators.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | assessed up to 1 years
  From the first time of treatment until the date of first documented progression or date of death from any cause, whichever comes first

SECONDARY OUTCOMES:
overall response rate (ORR) | assessed up to 2 years
  ORR is defined as the proportion of participants who have a partial response (PR) or complete response (CR) to therapy according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
overall survival (OS) | assessed up to 2 years
  OS is defined as the length of time from treatment to death from any cause
time to progression(TTP) | assessed up to 2 years
  From date of the first dose of study drug until the date of first documented progression NOT including death
duration of response (DOR) | assessed up to 2 years
  From the first date of response until the date of first documented progression

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Liu J, Yin R, Zou D, Zheng H, Cao J, Chen Z, Sun W, Gao Y, Zhang S, Zeng L, An R, Lu X, Ye S, Wu X. Efficacy and safety of chiauranib in a combination therapy in platinum-resistant or refractory ovarian cancer: a multicenter, open-label, phase Ib and II study. Mol Cancer. 2024 Aug 9;23(1):162. doi: 10.1186/s12943-024-02076-x. PMID 39123210